CLINICAL TRIAL: NCT00167895
Title: The Use of Platelet Derived Growth Factors in Total Knee Arthroplasty, a Randomized Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Westfries Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: M04-035
Record Dates: First submitted 2005-09-10; First posted 2005-09-14 (Estimated); Last update posted 2007-04-25 (Estimated); Status verified 2007-04

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; knee; platelet concentrate
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Adding platelet concentrate to the wound

SUMMARY:
The objective of this study is to evaluate the effect of autologous platelet concentrate on blood loss (post-operative decrease of haemoglobin concentration), wound healing complications, range of motion, pain reduction and outcome scores when used in total knee arthroplasty.

DETAILED DESCRIPTION:
The short-term functional recovery after a total knee arthroplasty (TKA) is largely dependent on initial wound healing. Haematoma formation may lead to prolonged wound drainage and tissue necrosis1, which can have a negative effect on early range of motion, post-operative pain and length of hospital stay. In addition, studies have suggested that prolonged wound drainage also leads to a higher infection rate.

To decrease haematoma formation, primary soft tissue homeostasis and adequate tissue repair are essential. During the immediate reaction of tissue to injury, haemostasis and inflammation occur. Growth factors, especially PDGF (platelet derived growth factor) and TGF-β (transforming growth factor-beta), play a crucial role in the biochemical cascade at the site of repair. These growth factors are mostly derived from platelets. They act as chemotactic agents for polymorphonuclear leucocytes, macrophages, fibroblasts and lymphocytes. Both factors stimulate angiogenesis and fibroplasia. PDGF also has a role in wound contraction and remodeling. When applying large concentrations of growth factors in a wound, faster tissue repair and homeostasis can be expected, thus leading to less haematoma formation.

Treatment with autologous platelet concentrate involves direct application of concentrated platelets, growth factors and fibrin in the operation wound. A small volume (55-110 ml) of the patient's own blood is taken to derive a platelet rich gel which can be sprayed directly into the wound.

The objective of this study is to evaluate the effect of autologous platelet concentrate on blood loss (post-operative decrease of haemoglobin concentration), wound healing complications, range of motion, pain reduction and outcome scores when used in total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary total knee arthroplasty for primary osteoarthritis

Exclusion Criteria:

* Coagulation disorder
* Abnormal pre-operative levels of APTT, PT and/or thrombocytes
* Homologous blood transfusion last 4 weeks
* Coagulation disorder
* Use of anticoagulation medication
* Use of any iron supplements or erythropoietin at time of operation or during 1 week prior to operation
* Primary bone tumor or metastatic bone disease
* Unable or unwilling to participate in follow-up
* Unable to give informed consent
* Previous infection in knee
* Use of corticosteroids at time of operation or during 4 weeks prior to operation
* Any neuromuscular disorder
* Active infection or osteomyelitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Decrease in post-operative blood haemoglobin concentration (as a measure for blood loss)
Number of days of wound drainage
Duration of hospital stay
Range of motion (ROM); flexion-extension using a goniometer

SECONDARY OUTCOMES:
Number of homologous blood packed cells needed after TKA
Pain score (VAS)
Wound complications
Amount and sort of analgesics required
Outcome scoring systems:
o International Knee Society TKA Score
o 12-questionnaire score
o SF-36
· Patient satisfaction using the Likert-scale

CONTACTS AND LOCATIONS:
Overall Officials: Karin S Peters, MD, Principal Investigator — Slotervaart Ziekenhuis
Locations (1):
- Westfries Gasthuis, Hoorn, Netherlands